CLINICAL TRIAL: NCT05850052
Title: Comparison of Comparison of McGrath Videolaryngoscopy and Direct Laryngoscopy for Rapid Sequence Intubation: an International, Multicenter Randomized Trial
Brief Title: McGrath Videolaryngoscopy and Direct Laryngoscopy Rapid Sequence Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: McGrady Study
Record Dates: First submitted 2023-04-25; First posted 2023-05-09 (Actual); Results first posted 2025-02-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- McGrath Videolaryngoscope for rapid endotracheal intubation (Experimental): The researchers will use the McGrath videolaryngoscope for rapid sequence endotracheal intubation.
  Interventions: Device: McGrath videolaryngoscope for rapid sequence endotracheal intubation
- Efficacy of conventional direct laryngoscopy (Other): The researchers seek to compare the efficacy of conventional direct laryngoscopy using a Macintosh blade.
  Interventions: Device: Conventional direct laryngoscopy using a Macintosh blade

INTERVENTIONS:
Device: McGrath videolaryngoscope for rapid sequence endotracheal intubation — Visualize a patient's airway to aid placement of tracheal tube with ease.
  Arms: McGrath Videolaryngoscope for rapid endotracheal intubation
Device: Conventional direct laryngoscopy using a Macintosh blade — Examine a patient's airway to aid placement of tracheal tube with ease.
  Arms: Efficacy of conventional direct laryngoscopy

SUMMARY:
The study seeks to compare the efficacy of conventional direct laryngoscopy using a Macintosh blade with the McGrath videolaryngoscope for rapid sequence endotracheal intubation.

DETAILED DESCRIPTION:
The study aims to conduct a multicenter international trial to enroll a maximum of 800 consenting adults who fall under the American Society of Anesthesiologists (ASA) physical status 1-3 category and require elective non-cardiac surgery necessitating endotracheal intubation with rapid sequence induction for general anesthesia. The study seeks to compare the efficacy of conventional direct laryngoscopy using a Macintosh blade with the McGrath videolaryngoscope for rapid sequence endotracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery requiring oral endotracheal intubation for general anesthesia;
* Anticipated extubation in the operating room;
* American Society of Anesthesiologists (ASA) physical status 2-3;
* Age between 18 and 99 years;
* Body Mass index ≥ 40 kg/m2.

Exclusion Criteria:

* Refusal of participation by attending anesthesiologist;
* Indicated rapid sequence induction for any reason including, but not limited to high risk of aspiration
* Indicated fiberoptic awake intubation.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2023-05-07 (Actual); Primary Completion 2024-06-05 (Actual); Study Completion 2024-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kurt Ruetzler, MD, Principal Investigator — The Cleveland Clinic
Locations (2):
- Turkey (Türkiye) (2):
  - The University of Health Science, Bakirkoy Dr. Sadi Konuk Education, and Research Hospital,, Istanbul
  - The University of Health Science, Konya City Hospital, Konya

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomization data were missing for n = 6 patients.
Groups:
- Efficacy of Conventional Direct Laryngoscopy: The researchers seeks to compare the efficacy of conventional direct laryngoscopy using a Macintosh blade,
  Conventional direct laryngoscopy using a Macintosh blade: Examine a patient's airway to aid placement of tracheal tube with ease.
Period: Overall Study
Arm/Group | McGrath Videolaryngoscope for Rapid Endotracheal Intubation | Efficacy of Conventional Direct Laryngoscopy
Started | 193 | 201
Completed | 193 | 201
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | McGrath Videolaryngoscope for Rapid Endotracheal Intubation | Efficacy of Conventional Direct Laryngoscopy | Total
Number analyzed (Participants) | 193 | 201 | 394
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 46 [35 to 56] | 46 [37 to 57] | 46 [36 to 57]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Gender data for one patient is missing in Direct laryngoscopy group
  Participants
    number analyzed (Participants) | 193 | 200 | 393
    Female | 119 | 109 | 228
    Male | 74 | 91 | 165
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Study center [Number; unit: participants]
  Istanbul | 96 | 104 | 200
  Konya | 97 | 97 | 194
BMI [Median (Inter-Quartile Range); unit: kg/m^2] | 28 [25 to 31] | 28 [25 to 31] | 28 [25 to 31]
History of difficult airway [Count of Participants; unit: Participants] — Population: This data for one patient is missing in Direct laryngoscopy group
  Participants
    Yes: number analyzed (Participants) | 193 | 200 | 393
    Yes | 6 | 7 | 13
    No: number analyzed (Participants) | 193 | 200 | 393
    No | 187 | 193 | 380
Mallampati score [Count of Participants; unit: Participants] — Population: The Mallampati score is missing for 1 patient in the McGrath Videolaryngoscope group and for 5 patients in the direct laryngoscopy group
  Participants
    I (Soft palate, uvula, pillars visible: number analyzed (Participants) | 192 | 196 | 388
    I (Soft palate, uvula, pillars visible | 59 | 54 | 113
    II (Soft palate, major part of uvula visible): number analyzed (Participants) | 192 | 196 | 388
    II (Soft palate, major part of uvula visible) | 89 | 104 | 193
    III (Soft palate, base of uvula visible): number analyzed (Participants) | 192 | 196 | 388
    III (Soft palate, base of uvula visible) | 39 | 35 | 74
    IV (Only hard palate visible: number analyzed (Participants) | 192 | 196 | 388
    IV (Only hard palate visible | 5 | 3 | 8
ASA physical status [Count of Participants; unit: Participants] — Population: This data for one patient is missing in Direct laryngoscopy group
  Participants
    1 (Healthy): number analyzed (Participants) | 193 | 200 | 393
    1 (Healthy) | 41 | 39 | 80
    2 (Mild systemic illness): number analyzed (Participants) | 193 | 200 | 393
    2 (Mild systemic illness) | 124 | 135 | 259
    3 (Severe systemic illness): number analyzed (Participants) | 193 | 200 | 393
    3 (Severe systemic illness) | 28 | 26 | 54

OUTCOME MEASURES:

1. Primary Outcome: Visualization of the Vocal Cords
Description: The visualization of the vocal cords, defined using the modified Cormack and Lehane classification:
  Grade I: Full view of the glottis (vocal cords are completely visible). Grade IIa: Partial view of the glottis (only the posterior portion of the glottis is visible).
  Grade IIb: Only the arytenoids or the posterior extremity of the vocal cords are visible (the anterior commissure is not seen).
  Grade III: Only the epiglottis is visible (the glottis is not visible). Grade IV: Neither the epiglottis nor the glottis is visible (only the soft palate is seen).
Time Frame: From the start time of intubation to time of the end of surgery, up to 12 hours.
Measure: Count of Participants; unit: Participants
Arm/Group | McGrath Videolaryngoscope for Rapid Endotracheal Intubation | Efficacy of Conventional Direct Laryngoscopy
Number analyzed (Participants) | 193 | 201
Participants
  Grade I - Full view of the glottis | 90 | 85
  Grade IIa - Partial view of the glottis | 63 | 67
  Grade IIb - Only the arytenoids or the posterior extremity of the vocal cords are visible | 26 | 28
  Grade III - Only the epiglottis is visible | 10 | 17
  Grade IV - Neither the epiglottis nor the glottis is visible | 4 | 4
Statistical Analysis 1: Comparison: McGrath Videolaryngoscope for Rapid Endotracheal Intubation vs Efficacy of Conventional Direct Laryngoscopy; Test type: Superiority; p = 0.26, proportional-odds cumulative logit model; Odds Ratio (OR) = 1.24, 95% CI 2-sided [0.85 to 1.79]

2. Secondary Outcome: Number of Participants With 1, 2, 3, and 4 Intubation Attempts
Description: An intubation attempt was recorded once the endotracheal tube entered the oral cavity
Time Frame: From the start time of intubation to time of the end of surgery, up to 12 hours.
Population: N = 4 patients were missing the number of attempts in the McGrath Videolaryngoscope group. N = 3 patients were missing the number of attempts in the Direct Laryngoscopy group.
Measure: Count of Participants; unit: Participants
Arm/Group | McGrath Videolaryngoscope for Rapid Endotracheal Intubation | Efficacy of Conventional Direct Laryngoscopy
Number analyzed (Participants) | 189 | 198
Participants
  1 intubation attempt | 167 | 176
  2 intubation attempts | 21 | 21
  3 intubation attempts | 0 | 1
  4 intubation attempts | 1 | 0
Statistical Analysis 1: Comparison: McGrath Videolaryngoscope for Rapid Endotracheal Intubation vs Efficacy of Conventional Direct Laryngoscopy; Test type: Superiority; p = 0.86, proportional-odds cumulative logit model; incidence rate ratio = 1.02, 97.5% CI 2-sided [0.82 to 1.27]

3. Secondary Outcome: Intubation Failure.
Description: Intubation was considered a failure if there was: (1) a failure to intubate after 3 attempts, (2) the need to switch intubators or intubation device, or (3) the need to stop study per anesthesiologist's discretion.
Time Frame: From the start time of intubation to time of the end of surgery, up to 12 hours.
Measure: Count of Participants; unit: Participants
Arm/Group | McGrath Videolaryngoscope for Rapid Endotracheal Intubation | Efficacy of Conventional Direct Laryngoscopy
Number analyzed (Participants) | 193 | 201
Participants | 3 | 1
Statistical Analysis 1: Comparison: McGrath Videolaryngoscope for Rapid Endotracheal Intubation vs Efficacy of Conventional Direct Laryngoscopy; Test type: Superiority; p = 0.36, Fisher Exact; Risk Ratio (RR) = 3.1, 95% CI 2-sided [0.32 to 30]

ADVERSE EVENTS:
Time Frame: From the start time of intubation to the end of the surgery, up to 12 hours.
Arm/Group | McGrath Videolaryngoscope for Rapid Endotracheal Intubation | Efficacy of Conventional Direct Laryngoscopy
All-Cause Mortality (participants affected / at risk) | 0/193 | 0/201
Serious Adverse Events (participants affected / at risk) | 0/193 | 0/201
Other Adverse Events (participants affected / at risk) | 0/193 | 0/201

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-24): https://cdn.clinicaltrials.gov/large-docs/52/NCT05850052/Prot_SAP_000.pdf